CLINICAL TRIAL: NCT05074199
Title: Comparison of Cosmetic Outcomes of Straight Line and W-plasty Techniques for Linear Wound Closure: a Randomized Evaluator Blinded Split Wound Comparative Effectiveness Trial
Brief Title: Comparison of Cosmetic Outcomes of Straight Line and W-plasty Techniques for Linear Wound Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1195990
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Suture Dermatologic; Surgery; Cosmetic Outcome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-plasty (Active Comparator): The cosmetic appearance of scars closed in a in a "zig-zag" " fashion (W-plasty).
  Interventions: Procedure: W-plasty/Linear closure
- Linear closure (Active Comparator): The cosmetic appearance of scars closed in a standard "straight line" fashion (linear closure).
  Interventions: Procedure: W-plasty/Linear closure

INTERVENTIONS:
Procedure: W-plasty/Linear closure — The patient's wound will be labeled A if it is on the left or superior side of the investigator and B if it is on the right or inferior side. A predetermined, concealed randomization number will be obtained from the RedCap randomization module, which will specify how side A is to be treated. Side B will be treated the opposite way as A. Side A will always be closed first. The side assigned to be closed in a traditional straight line (SL) will have the standing cutaneous deformity ("dog ear") excised in the standard manner using Burrow's triangles, resulting in an elliptical defect amenable to linear closure. The side assigned to be closed with W-plasty will have the dog ear excised in a zig-zag fashion consistent with the W plasty flap design. Both sides of the wound will receive subcuticular closure with interrupted subdermal sutures as is the standard of care, followed by a standard running cuticular closure with absorbable suture material.

SUMMARY:
The purpose of this study is to compare the cosmetic outcome of traditional straight-line (SL) linear closure to that of W plasty (a type of geometric broken-line cutaneous closure technique) for closure of post-auricular wounds resulting from harvest of full thickness skin grafts during Mohs micrographic surgery. The research team will use a split wound model, where half of the wound is repaired with a straight-line cutaneous closure and the other half is repaired with the W-plasty technique. Three-months post-surgery, the scar will be measured via the patient observer scar assessment scale (POSAS), a validated scar instrument. The scar width, and adverse events will also be recorded.

DETAILED DESCRIPTION:
Optimizing the cosmetic appearance of surgical scars is an important element of cutaneous surgery, especially for procedures performed on conspicuous areas of the body such as the head and face. Multiple factors have been shown to affect the aesthetic outcome of scars resulting from cutaneous surgery including the amount of tension on the resultant surgical wound, suture technique and type of sutures used. The use of various wound closure techniques including linear straight-line (SL) and geometric broken-line closure techniques (Z-plasty, W-plasty) to achieve a superior cosmetic scar outcome, has been debated in the dermatology and plastic surgery literature with few studies comparing SL and broken-line closure techniques and mixed results as to which modality provides a superior cosmetic outcome [2]. A study of forehead donor site closure in in 31 undergoing a paramedian forehead flap procedure showed that W-plasty provided a superior cosmetic outcome over straight-line closure, however another study in 30 patients undergoing tempo-parietal facial flaps found that W-plasty resulted in an inferior cosmetic outcome compared to linear closure. In addition, a large national survey of over 800 lay public participants found that linear scars were perceived as more cosmetically favorable than zig-zag scars in three facial locations (temple, cheek and forehead). Currently, there are no studies comparing the two closure techniques in a split-scar design, which can ameliorate many potentially confounding individual patient factors that could affect scar outcome.

Full-thickness skin grafts (FTSGs) are a commonly utilized reconstructive option in cutaneous surgery, and are typically harvested from behind the ear (postauricular) to close surgical defects on the head and face following surgical removal of both benign and malignant cutaneous tumors. This study aims to investigate whether the choice of straight-line linear closure versus a zig-zag broken line cutaneous closure technique (W-plasty) affects the cosmetic outcome of postauricular scars resulting from donor site closure following FTSG harvest. Additionally, skin lesions removed behind the ear present another opportunity to compare outcomes of these two techniques in an inconspicuous location.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head or face for which a full thickness skin graft will be used as part of the reconstruction or has a lesion that will be excised in mastoid area of the neck, behind the ear.
* Willing to return for follow up visit.

Exclusion Criteria:

* Wounds predicted to be less than 3 cm in size after closure.
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Patient Observer Scar Assessment Scale (POSAS) scores | 3-12 months
  The primary outcome is the difference in Patient Observer Scar Assessment Scale (POSAS) scores between the halves of the wound (standard linear closure versus W-plasty). The POSAS instrument incorporates separate questionnaires for observers and patients. Each questionnaire contains six items with possible scores from 0-10 for a total maximum score of 60 on each component (patient and observer).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehrzad M, Kang AS, Armstrong AW, Eisen DB. Comparing Cosmetic Outcomes of Straight-Line Versus W-Plasty Techniques for Linear Postauricular Wound Closure: A Randomized Evaluator Blind Split-Scar Trial. Dermatol Surg. 2024 May 1;50(5):423-427. doi: 10.1097/DSS.0000000000004113. Epub 2024 Feb 28. PMID 38416811